CLINICAL TRIAL: NCT06465641
Title: Effectiveness of Methylphenidate in Children and Adolescents With KBG Syndrome: An N-of-1 Series
Brief Title: Methylphenidate in KBG Syndrome: N-of-1 Series
Acronym: KBGS_N_of_1
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 113883
Record Dates: First submitted 2024-02-06; First posted 2024-06-20 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-02

CONDITIONS: Kbg Syndrome; ADHD - Combined Type
MeSH Terms: conditions — KBG syndrome | interventions — Methylphenidate

STUDY DESIGN:
Intervention Model Description: N-of-1 series (aggregated N-of-1 trial)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Methylphenidate (Active Comparator): Methylphenidate hydrochloride in capsules
  Interventions: Drug: Methylphenidate Hydrochloride
- Placebo (Placebo Comparator): Microcrystalline cellulose in capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylphenidate Hydrochloride — Methylphenidate hydrochloride in capsules
  Arms: Methylphenidate
Drug: Placebo — Microcrystalline cellulose in capsules
  Arms: Placebo

SUMMARY:
The goal of this clinical trial] is to learn about the effect of methylphenidate in children and adolescents with KBG syndrome. The main question it aims to answer is:

• What is the effectiveness of methylphenidate on attention deficit and ADHD-related symptoms in children and adolescents with KBG syndrome?

Participants will receive multiple blocks of treatment with methylphenidate and placebo and fill out various questionnaires.

DETAILED DESCRIPTION:
KBG syndrome (KBGS) is a neurodevelopmental disorder (NDD) characterized by developmental delay and/or intellectual disability, typical facial features, skeletal and congenital anomalies.

Behavioural issues are a frequent feature, reported in 50-94% of persons with KBGS.The behavioural problems are diverse, and include attention deficit hyperactivity disorder (ADHD), autism spectrum disorder (ASD), obsessive-compulsive disorder, anxiety, and difficulties in social situations. Van Dongen et al. systematically investigated the behavioural and cognitive phenotype of KBGS patients. This study showed a high level of distractibility, impulsivity and restless behaviour in KBGS patients. As a tertiary reference centre for KBGS in the Netherlands, the investigators notice there is an unmet need for evidence-based interventions for the behavioral problems related to KBGS. A previous survey amongst KBGS caretakers confirmed that (features of) attention-deficit/hyperactivity disorder (ADHD) are the most frequently reported behavioural problems in children with KBGS. Furthermore, the study results indicate that methylphenidate (MPH) has a good effect on ADHD-related symptoms in KBGS, as this is reported by most parents. The promising results from this first exploration on MPH in KBGS indicate that it seems even more effective than in the general population of children with ADHD. However, evidence-based data on optimal dosing and adverse events are lacking. Remarkably, only 2/12 KBGS patients who were treated with stimulants such as MPH had an official ADHD diagnosis. This indicates that patients with ADHD-related symptoms fitting with a probability diagnosis of ADHD, but who do not necessarily fit all the Diagnostic and statistical manual 5 (DSM-5) criteria for ADHD, may also benefit from drug treatment.

The investigators will examine the effectiveness of MPH in children and adolescents with KBGS and (a probability diagnosis of) ADHD, using an N-of-1 series (aggregated N-of-1) trial design.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-20 years
* Molecularly confirmed diagnosis of KBG syndrome (pathogenic ANKRD11 variant or a chromosome 16q24 deletion including ANKRD11)
* Attention deficit or ADHD-related symptoms or a formal ADHD diagnosis, with a significant impact on daily life*
* Presence of a subject's caregiver or supervisor for proxy-reports

Exclusion Criteria:

* Family history of acute cardiac death that warrants further cardiac investigation
* Cardiovascular disease in medical history (severe hypertension, heart failure, arterial occlusive disease, potentially life-threatening arrythmias, angina pectoris, hemodynamically significant congenital heart defect, cardiomyopathy, myocardial infarction and channelopathy)
* Current or previous presence of hyperthyroidism, glaucoma or pheochromocytoma
* Use of (psychotropic/stimulant) drugs which interact with MPH
* Schizophrenic or psychotic disorder in medical history
* Unstable epilepsy (not controlled with medication)
* History of frequent drug and/or alcohol abuse
* Excessive alcohol/drug use and/or intoxication with one or both during the study
* Pregnant or lactating women
* Inability to understand or speak Dutch

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Strenghts and difficulties questionnaire, ADHD subscale | Baseline, and daily in week 1,3,5,7,9,11
  Minimum score 1, maximum score 10 (higher score is worse outcome).

SECONDARY OUTCOMES:
Strenghts and difficulties questionnaire, emotional problems subscale | Baseline, and daily in week 1,3,5,7,9,11
  Minimum score 1, maximum score 10 (higher score is worse outcome).
Dutch shortened version of the Emotion Dysregulation Inventory (EDI) reactivity index | Baseline, and daily in week 1,3,5,7,9,11
  Minimum score 0, maximum score 28 (higher score is worse outcome)
Goal Attainment Scoring (GAS) | Baseline, and at the end of week 1,3,5,7,9,11
  Personal goals, no minimum or maximum score
Personal Questionnaire (PQ) | Baseline, and at the end of week 1,3,5,7,9,11
  Personal goals, no minimum or maximum score
Adverse Effects checklist for methylphenidate | Baseline, and daily in week 1,3,5,7,9,11
  Checklist of adverse effects
McMaster Family assessment device (FAD), subscale General Functioning | Baseline, and at the end of week 1,3,5,7,9,11
  10 items, 4 point scale, maximum score 40
Autism diagnostic observation scale (ADOS-2) | Baseline
  Minimum score 15, maximum score 60 (cut-off score for autism is 30)

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University Medical Center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Individual patients data that underlie the results after deidentification, study protocol, and statistical analysis plan will be shared upon request following publication, to researchers who provide a methodologically sound proposal.
Supporting Information: Study Protocol, SAP
Time Frame: After publication, no end date
Access Criteria: Researchers who provide a methodologically sound proposal.